CLINICAL TRIAL: NCT04465188
Title: Scleral Buckling for Retinal Detachment Prevention in Genetically Confirmed Stickler Syndrome : a Randomized Controlled Trial
Brief Title: Scleral Buckling for Retinal Detachment Prevention in Genetically Confirmed Stickler Syndrome
Acronym: STL-DR-PREV
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P160948J; 2018-A01081-54 (Other: ID-RCB)
Record Dates: First submitted 2020-07-08; First posted 2020-07-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Stickler Syndrome
Keywords: Stickler syndrome; Retinal detachment; Prophylaxis; Collagen
MeSH Terms: conditions — Stickler syndrome, type 1; Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Surgical procedure to prevent retinal detachment in the unaffected eye
  Interventions: Procedure: Encircling scleral buckle surgical procedure
- Control arm (No Intervention): Standard procedure of clinical practice without any surgical procedure for the unaffected fellow eye.

INTERVENTIONS:
Procedure: Encircling scleral buckle surgical procedure — Encircling scleral buckle surgical procedure under general anesthesia
  Arms: Experimental arm

SUMMARY:
The purpose of this study is to determine whether a scleral buckling surgical procedure performed on fellow eyes of patients with genetically confirmed Stickler syndrome can prevent the occurrence retinal detachment and/or severe vision loss of the study eye.

DETAILED DESCRIPTION:
Stickler syndrome (STL) is a genetic disease affecting several organs. However the major risk is represented by the development of retinal detachment (RD). Up to 80% of patients present a RD and 25% to 80% have sequential bilateral RD. The surgical outcome of RD in this population is worse than that of the general RD population mainly because of the severity at diagnosis and the high frequency and severity of postoperative complications. Prevention has therefore emerged as a therapeutic option for this identifiable high-risk group of patients. Prevention has been proposed especially for the fellow (contralateral) eye of patients having presented a RD in their first eye and often lost vision as a consequence of retinal detachment in the first eye.

The investigators hypothesize that a scleral buckling surgical procedure performed for the fellow eye of STL patients having recently presented a RD of the first eye could prevent the occurrence of bilateral RD and/or vision loss.

Stickler patients are regularly diagnosed and followed-up in referral centers mainly in the context of a recent retinal detachment. They are proposed genetic testing as part of the standard of care. Genetically confirmed Stickler patients having recently presented (<24 months) a retinal detachment and treated as part of the standard care are eligible for this study. During the usual follow-up visits performed for their recent first RD operation they will be informed and offered to participate in the "STL-DR-PREV study" for the prevention of RD of their fellow eye.

Patients in the intervention arm will undergo an encircling scleral buckle surgical procedure, which is a routine surgical procedure used for decades and still in use to treat RD that will be performed in the present study to prevent rather than to treat retinal detachment from a healthy eye of a patient having a genetically confirmed Stickler Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed Stickler Syndrome
* Aged 5 to 35
* Recent retinal detachment in the non-study eye (<24 months)
* Signed informed consent to participate in the study
* Sufficient patient cooperation to perform a complete ophthalmologic examination including a dilated fundus examination

Exclusion Criteria:

* Any type of previous prevention (laser, cryotherapy, scleral buckle) for the study eye
* Subclinical retinal rhegmatogenous detachment in the study eye.
* Any other ocular disease unrelated to Stickler syndrome significantly affecting visual acuity (ETDRS BCVA<20/400).
* Contraindications to general anesthesia
* Posterior vitreoretinal traction on optical coherence tomography
* Intraoperative detection of one or more of the above-mentioned non-inclusion criteria

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity and retinal detachment rate | 5 years
  Early Treatment Diabetic Retinopathy Study (ETRDS) best corrected visual acuity (BCVA) and dilated funduscopic examinations at scheduled follow-up (every 6 months)

SECONDARY OUTCOMES:
Rate of retinal breaks | 5 years
Rate of intravitreal hemorrhage | 5 years
Outcome in prevention-failed study eyes | 5 years
  outcome of surgery for RD in the study eye of patients for whom prevention failed and had to be operated on for RD repair of the study eye
Effect of add-on cryotherapy | 5 years
  To assess within the experimental arm whether patients having had cryotherapy as part (allowed by the protocol at the surgeon's discretion in addition to the standard procedure) of the scleral buckling procedure present a decrease in the rate of RD as compared to buckled patients without cryotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BREZIN, MD,Phd, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monin C, Van Effenterre G, Andre-Sereys P, Haut J. [Prevention of retinal detachment in Wagner-Stickler disease. Comparative study of different methods. Apropos of 22 cases]. J Fr Ophtalmol. 1994;17(3):167-74. French. PMID 8182253
- [Background] Abeysiri P, Bunce C, da Cruz L. Outcomes of surgery for retinal detachment in patients with Stickler syndrome: a comparison of two sequential 20-year cohorts. Graefes Arch Clin Exp Ophthalmol. 2007 Nov;245(11):1633-8. doi: 10.1007/s00417-007-0609-2. Epub 2007 Jun 20. PMID 17579881
- [Background] Carroll C, Papaioannou D, Rees A, Kaltenthaler E. The clinical effectiveness and safety of prophylactic retinal interventions to reduce the risk of retinal detachment and subsequent vision loss in adults and children with Stickler syndrome: a systematic review. Health Technol Assess. 2011 Apr;15(16):iii-xiv, 1-62. doi: 10.3310/hta15160. PMID 21466760
- [Background] Ang A, Poulson AV, Goodburn SF, Richards AJ, Scott JD, Snead MP. Retinal detachment and prophylaxis in type 1 Stickler syndrome. Ophthalmology. 2008 Jan;115(1):164-8. doi: 10.1016/j.ophtha.2007.03.059. Epub 2007 Aug 2. PMID 17675240
- [Background] Fincham GS, Pasea L, Carroll C, McNinch AM, Poulson AV, Richards AJ, Scott JD, Snead MP. Prevention of retinal detachment in Stickler syndrome: the Cambridge prophylactic cryotherapy protocol. Ophthalmology. 2014 Aug;121(8):1588-97. doi: 10.1016/j.ophtha.2014.02.022. Epub 2014 May 1. PMID 24793526